CLINICAL TRIAL: NCT05593575
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Parallel, Dose-finding Phase 2 Clinical Study to Evaluate the Efficacy and Safety of SPH3127 Tablets in the Treatment of Diabetic Kidney Disease
Brief Title: Efficacy and Safety of SPH3127 Tablets on Treating the Diabetic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPH3127-202
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SPH3127-1 (Experimental): 1 tablet of SPH3127 (50 mg) ，3 tablets of SPH3127 (50mg)matching placebo， 1 capsule of valsartan matching placebo, orally, once daily for 12 consecutive weeks
  Interventions: Drug: SPH3127+SPH3127matching placebo+valsartan matching placebo
- SPH3127-2 (Experimental): 2 tablet of SPH3127 (50 mg) ，2 tablets of SPH3127 (50mg)matching placebo， 1 capsule of valsartan matching placebo, orally, once daily for 12 consecutive weeks
  Interventions: Drug: SPH3127+SPH3127matching placebo+valsartan matching placebo
- SPH3127-3 (Experimental): 4 tablet of SPH3127 (50 mg) ，1 capsule of valsartan matching placebo, orally, once daily for 12 consecutive weeks
  Interventions: Drug: SPH3127+valsartan matching placebo
- SPH3127-4 (Experimental): 4 tablets of SPH3127 (50mg)matching placebo， 1 capsule of valsartan , orally, once daily for 12 consecutive weeks
  Interventions: Drug: SPH3127 matching placebo+valsartan

INTERVENTIONS:
Drug: SPH3127+SPH3127matching placebo+valsartan matching placebo — 1 tablet of SPH3127 (50 mg) ，3 tablets of SPH3127 (50mg)matching placebo， 1 capsule of valsartan matching placebo, orally, once daily for 12 consecutive weeks
  Arms: SPH3127-1
Drug: SPH3127+SPH3127matching placebo+valsartan matching placebo — 2 tablet of SPH3127 (50 mg) ，2 tablets of SPH3127 (50mg)matching placebo， 1 capsule of valsartan matching placebo, orally, once daily for 12 consecutive weeks
  Arms: SPH3127-2
Drug: SPH3127+valsartan matching placebo — 4 tablet of SPH3127 (50 mg) ， 1 capsule of valsartan matching placebo, orally, once daily for 12 consecutive weeks
  Arms: SPH3127-3
Drug: SPH3127 matching placebo+valsartan — 4 tablets of SPH3127 (50mg)matching placebo， 1 capsule of valsartan, orally, once daily for 12 consecutive weeks
  Arms: SPH3127-4

SUMMARY:
To preliminarily evaluate the efficacy and safety of the renin inhibitor (SPH3127 tablets) in reduction in proteinuria in patients with diabetic kidney disease with valsartan as the comparator, and determine the recommended dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are diagnosed with type 2 diabetes who have been treated with at least one hypoglycemic therapy within 12 months prior to screening, with basically stable blood glucose level during screening;
2. During screening period, 120 mmHg ≤ sitting SBP ≤ 160 mmHg and sitting DBP < 110 mmHg;
3. Laboratory results before randomization should be: 1) at least twice the result of UCAR should be 30 mg/g ≤ UACR < 3000mg/g at W-8, W-4, W-2, and W0; 2) EGFR ≥ 45mL/min/1.73 m2 at W-4 and W0; 3) AST and ALT ≤ 2 times the upper limit of normal (ULN), and total bilirubin ≤ 1.5 times ULN at W0; 4) hemoglobin ≥ 90 g/L at W0; 5) 3.5 mmol/L ≤Serum potassium ≤ 4.8 mmol/L at W-4 and W0;
4. Subjects who agree to take effective contraceptive measures with their spouses throughout the study period and for up to 12 weeks after the last dose;
5. Subjects who thoroughly learn about the nature, significance, possible benefits, possible inconvenience and potential risks of the trial, and understand the study procedures and voluntarily sign the informed consent form prior to their participation in the trial.

Exclusion Criteria:

1. Sitting SBP >140 mmHg and/or sitting DBP >90 mmHg at baseline (W0);
2. Color ultrasonography of renal artery indicated renal artery stenosis;
3. ① Acute renal insufficiency② acute nephritic syndrome, polycystic kidney, kidney stone, nephrotic syndrome; ③there is evidence that proteinuria originates from primary and secondary renal diseases other than hypertensive renal damage; ④ gross hematuria in the past one year.
4. During the screening/run-in period, major modifications need to be made to the subject's corresponding treatment regimen due to poor control of other underlying diseases based on the investigator's judgement;
5. Subjects with fundus lesions in malignant hypertensive, such as retinal hemorrhage and papilledema;
6. Subjects who need to continuously take glucocorticoids, anti-tumor chemical or biological agents, and non-steroidal anti-inflammatory drugs during the study period;
7. Subjects with a history of acute myocardial infarction, coronary artery revascularization, Class IV heart failure, acute cerebral infarction, cerebral hemorrhage and transient ischemic attack within 3 months prior to randomization;
8. Subjects who have abnormal thyroid function tests with clinically significance;
9. Subjects with poor control of diabetes: HbA1c ≥ 9.0% at W0;
10. Subjects who have undergone major surgery within 3 months prior to screening or need to undergo major surgery during the trial;
11. Subjects whose medication adherence in the run-in period is < 80% or > 120%;
12. Subjects with a history of gastrointestinal surgery that may significantly change the absorption, distribution, metabolism and excretion of drugs;
13. Subjects who are known to be allergic to renin inhibitors, ARBs, ACEIs and their excipients, or those with hypersensitive constitution, or those who experience serious adverse reactions;
14. Women during pregnancy or lactating;
15. Subjects who need transplantation before randomization and during the trial;
16. Subjects with HIV infection, hepatitis B infection, hepatitis C infection, or other active infections;
17. Subjects who have a history of malignant tumor, and those who are suspected of malignant tumor;
18. Subjects with a past and current history of mental illness;
19. Subjects with a history of drug abuse or alcohol abuse within 2 years prior to screening;
20. Subjects who have participated in clinical trials of other drugs/devices as a subject within 3 months prior to screening;
21. Subjects with other diseases or conditions that the investigator considers not suitable for this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in UACR | at the end of Week 12 of treatment
  Percentage change from baseline in log-transformed UACR at the end of Week 12 of treatment

SECONDARY OUTCOMES:
Percentage change from baseline in UACR | at the end of Weeks 2, 4 and 8 of treatment
  Percentage change from baseline in log-transformed UACR at the end of Weeks 2, 4 and 8 of treatment
Percentage change from baseline in UPCR | at the end of Weeks 2, 4, 8 and 12 of treatment
  Percentage change from baseline in log-transformed UPCR at the end of Weeks 2, 4, 8 and 12 of treatment
The change trend of eGFR | from baseline to the end of Weeks 2, 4, 8 and 12 of treatment
  The change trend of eGFR from baseline to the end of Weeks 2, 4, 8 and 12 of treatment

CONTACTS AND LOCATIONS:
Locations (45):
- China (45):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The 900 Hospital of the Joint Service Support Force of the People's Liberation Army of China, Fuzhou, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital，Sun Yat sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Harbin Medical University Affiliated Fourth Hospital, Harbin, Heilongjiang
  - Luoyang Third People's Hospital, Luoyang, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Third Hospital of Wuhan, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Norman Bethune Hospital of Jilin University, Changchun, Jilin
  - The First People's Hospital of Yinchuan, Yinchuan, Ningxia
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - Xi'an Daxing Hospital, Xi’an, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Zigong Fourth People's Hospital, Zigong, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Taizhou Municipal Hospital, Taizhou, Zhejiang
  - Beijing Tsinghua Changgeng Hospital, Beijin
  - Beijing Anzhen Hospital，Capital Medical University, Beijing
  - Beijing Tiantan Hospital，Capital Medical University, Beijing
  - Beijing Tongren Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Xiangya Hospital Central South University, Changsha
  - Chengdu Seventh People's Hospital, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital of Sichuan University, Chengdu
  - Shunde Hospital of Southern Medical University, Foshan
  - The Second Affiliated Hospital of Hainan Medical University, Haikou
  - Huizhou First Hospital, Huizhou
  - Qilu Hospital of Shandong University, Jinan
  - The First Affiliated Hospital of Shandong First Medical University, Jinan
  - Ningbo No.2 Hospital, Ningbo
  - Affiliated Zhongshan Hospital of Fudan University，Qingpu Branch, Shanghai
  - Ruijin Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Fengxian District Central Hospital, Shanghai
  - Shanghai Minhang District Central Hospital, Shanghai
  - Sheng Jing Hospital of China Medical University, Shenyang
  - The First Affiliated Hospital of China Medical University, Shenyang
  - The Seventh Affiliated Hospital，Sun Yat-sen University, Shenzhen
  - Second Hospital of Shanxi Medical University, Taiyuan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786